CLINICAL TRIAL: NCT04666207
Title: A Cohort Study of Non-hospitalized SARS-CoV-2 Positive Children in Denmark: Viral Shedding, Symptoms and Exposure
Brief Title: Viral Shedding, Symptoms and Exposure of SARS-CoV-2 in Non-hospitalized Children With COVID-19
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Allan Bybeck Nielsen, Dr., Rigshospitalet, Denmark
Other Study IDs: H-20028631-1
Record Dates: First submitted 2020-11-08; First posted 2020-12-14 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — feces, saliva, nasal secretions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR — RT-PCR for SARS-CoV-2

SUMMARY:
Data on COVID-19 in children are still scarce, and their role in SARS-CoV-2 transmission is poorly described. Furthermore, documentation of the best SARS-CoV-2 sampling methods in children are limited. In adults, saliva seems like a promising specimen to collect by noninvasive procedure to diagnose and monitor viral load of SARS-CoV-2, but this has not been tested in children yet.

We want to test the following hypothesis:

1. Shedding load and duration of SARS-CoV-2 in children are related to age, gender, clinical symptoms and exposure
2. Salvia samples have equal or higher sensibility than nasal swaps in children for detection of SARS-CoV-2
3. Parental home testing of saliva and feces is feasible in children

The study is a prospective cohort study of SARS-CoV-2 PCR-positive children from two test centers in the Capital Region of Denmark. Children aged 0-17 years with a PCR-positive SARS-CoV-2 test from a nasal or pharyngeal swab is included from May 2020 to January 2021 and followed-up for a period of 28 days with weekly sample collection and questionnaires.

Samples include a saliva sample, a nasal swap and a rectal swap for children under four years of age. A semiquantitative RT-PCR method, will identify positive and negative samples and provide a Ct value estimating viral load. Saliva and fecal samples will be analyzed from November 2020-February 2021.

Shedding duration will be related to medial history, clinical presentation, exposure, gender and age.

ELIGIBILITY:
Inclusion Criteria:

* a PCR-positive SARS-CoV-2 test

Exclusion Criteria:

-

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: SARS-CoV-2 PCR-positive children from two test centers in the Capital Region of Denmark
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Salvia samples have equal or higher sensibility than nasal swaps in children for detection of SARS-CoV-2 | 1 year
  Measured by RT-PCR

SECONDARY OUTCOMES:
Parental home testing of saliva and feces is feasible in children | 1 year
  measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ulrikka Nygaard, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen University Hospital Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No